CLINICAL TRIAL: NCT01388686
Title: Retrospective Analysis of Proven Bacteremia, CVC-associated Infections and Sepsis
Brief Title: Prevalence of CVC-associated Sepsis and Use of Blood Cultures in Berlin - Brandenburg
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Prof. MD, Director of the Dept. of Anaesthesiology and Intensive Care Medicine, CVK, CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: BAC_BLOOD
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Bacteremia
Keywords: sepsis; catheter; blood stream infection; blood culture
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INABBRA: Participating intensive care units of hospitals in the INABBRA alliance.

SUMMARY:
Structured web-based survey in selected hospitals with intensive care units in Berlin- Brandenburg to collect data on the overall number of blood cultures (used) and the prevalence of (positive blood cultures in patients with) CVC - associated sepsis.

DETAILED DESCRIPTION:
The use of CVC represents one of the major risk factors for sepsis, a highly prevalent disease in ICUs. Blood cultures obtained prior to antibiotic administration are part of the SSC Resuscitation Bundle and essential for the outcome of the patient. The CDC criteria to diagnose sepsis do not take into account the overall number of blood cultures obtained and thus, lead to an underestimation of the true incidence of sepsis. Up to now, few data is available on the total number of blood cultures obtained and the relation to the incidence of sepsis in German ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care units of hospitals in the INABBRA alliance.
* Patients with bacteremia.

Exclusion Criteria:

* Hospitals without intensive care unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bacteremia on intensive care units of different primary and secondary care hospitals in the region of Berlin-Brandenburg.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Total number of blood cultures drawn and total number of positive findings in ICUs | 1 year
  Retrospective analysis of cases with positive bloodculture among patients in ICU setting compared to the total amount of blood cultures taken in the same period of time and same hospital.

SECONDARY OUTCOMES:
Prevalence on CVC - associated sepsis/CLABSIs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Brun-Buisson C, Doyon F, Carlet J. Bacteremia and severe sepsis in adults: a multicenter prospective survey in ICUs and wards of 24 hospitals. French Bacteremia-Sepsis Study Group. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):617-24. doi: 10.1164/ajrccm.154.3.8810595.
- [Background] Tacconelli E, Smith G, Hieke K, Lafuma A, Bastide P. Epidemiology, medical outcomes and costs of catheter-related bloodstream infections in intensive care units of four European countries: literature- and registry-based estimates. J Hosp Infect. 2009 Jun;72(2):97-103. doi: 10.1016/j.jhin.2008.12.012. Epub 2009 Feb 25. PMID 19246122
- [Background] Brun-Buisson C, Doyon F, Carlet J, Dellamonica P, Gouin F, Lepoutre A, Mercier JC, Offenstadt G, Regnier B. Incidence, risk factors, and outcome of severe sepsis and septic shock in adults. A multicenter prospective study in intensive care units. French ICU Group for Severe Sepsis. JAMA. 1995 Sep 27;274(12):968-74. PMID 7674528
- [Background] Gastmeier P, Geffers C. [Nosocomial infections in Germany. What are the numbers, based on the estimates for 2006?]. Dtsch Med Wochenschr. 2008 May;133(21):1111-5. doi: 10.1055/s-2008-1077224. German. PMID 18478503
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710